CLINICAL TRIAL: NCT04912440
Title: Motorized Spiral Enteroscopy-assisted ERCP in Surgically Altered Anatomy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Evangelisches Krankenhaus Düsseldorf (Other)
Responsible Party: Sponsor
Other Study IDs: EVK-PSE-ERCP RETRO
Record Dates: First submitted 2021-05-28; First posted 2021-06-03 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Ercp in Altered Anatomy
Keywords: endoscopy; enteroscopy; ercp in altered anatomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MSE-ERCP: Group of patients, that received motorized spiral enteroscopy assisted ERCP in altered anatomy at the single study center
  Interventions: Device: MSE-ERCP

INTERVENTIONS:
Device: MSE-ERCP — No interventional study, MSE-ERCP performed within routine treatment, (approved indication of device)

SUMMARY:
Patients with surgically altered anatomy receiving Motorized Spiral Eneroscopy (MSE)-assisted ERCP at a single endoscopic reference center for various indications are planned to be retrospectively enrolled

DETAILED DESCRIPTION:
All consecutive patients with altered upper gastrointestinal anatomy after Billroth-II- or Roux-en-Y reconstructive surgery and indication for ERCP with biliary and/or pancreatic indication, who underwent routine Enteroscopy-assisted ERCP using MSE, at the study center during the study period, will be enrolled in the analysis.

Primary endpoint of the study will be efficacy and safety of MSE-assisted ERCP.

Retrospective epidemiologic Study (not interventional) was approved by local IRB and ethical committee of the North-Rhine Chamber of Physicians (Düsseldorf, Germany), Reference Number: 177/2021.

ELIGIBILITY:
Inclusion Criteria:

* altered upper gastrointestinal anatomy after Billroth-II- or Roux-en-Y reconstructive surgery
* indication for ERCP with biliary and/or pancreatic indication
* Enteroscopy-assisted ERCP using MSE, at the study center during the study period

Exclusion Criteria:

- due to the retrospective design of the study, no exclusion criteria are defined

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with surgically altered upper gastrointestinal anatomy and indication for endoscopic retrograde cholangio-pancreatography
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Success rate of MSE-ERCP | intraprocedural
  rate of subjects with successfull MSE-assisted ERCP
Adverse event rate of MSE-ERCP | 3 days
  rate of adverse events during and early after MSE-ERCP

SECONDARY OUTCOMES:
Success rate of enteroscopy | intraprocedural
  rate of subjects with successful enteroscopic access to the papilla
Procedural duration | intraprocedural
  overall time for MSE-ERCP (scope in to scope out)

CONTACTS AND LOCATIONS:
Overall Officials: Torsten Beyna, MD PhD, Principal Investigator — Evangelisches Krankenhaus Düsseldorf, Department of Gastroenterology and Therapeutic Endoscopy
Locations (1):
- Evangelisches Krankenhaus, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: No
No exchange of individual data is planned